CLINICAL TRIAL: NCT02399371
Title: A Phase II Study of the Anti-PD-1 Antibody Pembrolizumab in Patients With Malignant Mesothelioma
Brief Title: Pembrolizumab in Treating Patients With Malignant Mesothelioma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB14-1381; NCI-2015-00348 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IRB14-1381 (Other: University of Chicago Comprehensive Cancer Center); P30CA014599 (NIH)
Record Dates: First submitted 2015-03-13; First posted 2015-03-26 (Estimated); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Biphasic Mesothelioma; Epithelioid Mesothelioma; Peritoneal Malignant Mesothelioma; Pleural Biphasic Mesothelioma; Pleural Epithelioid Mesothelioma; Pleural Malignant Mesothelioma; Pleural Sarcomatoid Mesothelioma; Recurrent Peritoneal Malignant Mesothelioma; Recurrent Pleural Malignant Mesothelioma; Sarcomatoid Mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant; Solitary Fibrous Tumor, Pleural | interventions — pembrolizumab; Pharmacogenomic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (pembrolizumab) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 24 months in the absence of disease progression or unacceptable toxicity. Patients may be eligible for up to 1 year of additional pembrolizumab therapy if they progress after stopping pembrolizumab.
  Interventions: Biological: Pembrolizumab; Other: Laboratory Biomarker Analysis; Other: Pharmacogenomic Study

INTERVENTIONS:
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacogenomic Study — Correlative studies

SUMMARY:
This phase II trial studies how well pembrolizumab works in treating patients with malignant mesothelioma, a cancer of the linings around the lungs (pleura) or abdomen (peritoneum). Monoclonal antibodies, such as pembrolizumab, work by blocking a protein called programmed cell death 1 (PD-1) which may stimulate an immune response and kill tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the objective response rate of patients with malignant mesothelioma treated with pembrolizumab in A) an unselected patient population, as well as B) in a programmed cell death ligand 1 (PD-L1) positive population (should the trial proceed to Part B, and PD-L1 expression correlate with improved efficacy).

II. To determine the optimal threshold for PD-L1 expression using the 22C3 antibody based immunohistochemistry (IHC) assay in correlation to tumor response.

SECONDARY OBJECTIVES:

I. To determine the progression-free survival of patients with malignant mesothelioma in A) an unselected patient population and B) a PD-L1 positive population when treated with pembrolizumab.

II. To determine the overall survival of patients with malignant mesothelioma in A) an unselected patient population and B) a PD-L1 positive population when treated with pembrolizumab.

III. To determine the disease control rate (complete response [CR] + partial response [PR] + stable disease [SD]) of patients with malignant mesothelioma who are treated with pembrolizumab in A) an unselected patient population and B) a PD-L1 positive population.

IV. To determine toxicity in patients with malignant mesothelioma who are treated with pembrolizumab.

V. To determine percentage of patients with mesothelioma who have PD-L1 tumor expression, and the distribution of PD-L1 expression (percent positivity of tumor cells/stroma staining).

TERTIARY OBJECTIVES:

I. To characterize the T-cell inflamed phenotype in mesothelioma patients via presence of cluster of differentiation (CD)8 tumor infiltrating lymphocytes (TILs) and/or use of a gene expression signature (Nanostring).

II. To evaluate other immune escape mechanisms including indoleamine-pyrrole 2,3-dioxygenase (IDO) expression, regulatory T cells (Tregs) (forkhead box P3 [FOXP3] expression), myeloid-derived suppressor cells (MDSCs) and other checkpoints by immunohistochemistry (or other methods e.g. flow cytometry).

III. To determine PD-L1 expression by mass spectrometry and correlate with tumor response, PD-L1 expression by IHC, and the T-cell inflamed phenotype.

IV. To determine the immune cell populations present in fresh tumor (when available), via tumor digests and mass spectrometry-based flow cytometric analysis (e.g. using CyTOF) in a multiplex fashion in patients with fresh tumor tissue.

V. To characterize the T-cell receptor repertoire of TILs compared to circulating T-cells in mesothelioma patients with available fresh frozen tissue (spectrotyping, T-cell repertoire sequencing [e.g. using the Adaptive platform]).

OUTLINE:

Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1. Treatment repeats every 21 days for up to 24 months in the absence of disease progression or unacceptable toxicity. Patients may be eligible for up to 1 year of additional pembrolizumab therapy if they progress after stopping pembrolizumab.

After completion of study treatment, patients are followed up for 30 days (up to 90 days for serious adverse events), every 8 weeks until patient experiences confirmed disease progression or starts a new anti-cancer therapy, and then every 12 weeks for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed pleural or peritoneal malignant mesothelioma, epithelial, sarcomatoid, or biphasic subtypes
* Disease progression on or after pemetrexed and cis- or carboplatin
* ONLY FOR PART B - PD-L1 selection should a PD-L1 expression threshold have been defined in Part A and potentially additional mesothelioma trial data; there will be no PD-L1/biomarker selection for Part A
* No more than 2 prior lines of cytotoxic therapy, which should have included pemetrexed and a platinum
* Enrollment of treatment naïve patients who refuse standard chemotherapy or are intolerant may be permissible if reviewed and deemed clinically appropriate by the principal investigator (PI)
* Be willing and able to provide written informed consent for the trial
* Have measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 for peritoneal mesothelioma, and modified RECIST for pleural mesothelioma
* Have provided tissue from an archival tissue sample or newly obtained core or excisional biopsy of a tumor lesion; while 20 unstained slides or a tumor block are preferred, at least 14 unstained slides are requested for analysis; PI approval for a lower number of slides is acceptable
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) performance scale
* Absolute neutrophil count (ANC) >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 9 g/dL
* Serum creatinine =< 1.5 X upper limit of normal (ULN) OR measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) >= 50 mL/min for subject with creatinine levels > 1.5 X institutional ULN; creatinine clearance should be calculated per institutional standard
* Serum total bilirubin =< 1.5 X ULN OR direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 ULN
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X ULN OR =< 5 X ULN for subjects with liver metastases
* International normalized ratio (INR) or prothrombin time (PT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants
* Activated partial thromboplastin time (aPTT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Female subjects of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication; if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication; subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy

Exclusion Criteria:

* Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 2 weeks (4 weeks for monoclonal antibodies) of the first dose of treatment
* Side effects from prior treatment have not resolved to =< grade 1 (or baseline due to previously administered agent/pre-existing conditions)
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment
* Has had a prior monoclonal antibody within 4 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to a previously administered agent

  * Note: Subjects with =< grade 2 neuropathy are an exception to this criterion and may qualify for the study
  * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Has a known additional malignancy that is progressing or requires active treatment; exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, in situ cervical cancer, or other indolent cancers which either have undergone curative-intent therapy or inactive (i.e. not expected to limit life expectancy or interfere with therapy)
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis; subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment
* Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents; subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule; subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study; subjects with hypothyroidism stable on hormone replacement or Sjorgen's syndrome will not be excluded from the study
* Has evidence of interstitial lung disease or active, non-infectious pneumonitis
* Has an active infection requiring systemic therapy
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
* Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways)
* Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
* Has known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected)
* Has received a live vaccine within 30 days prior to the first dose of trial treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2015-03-31 (Actual); Primary Completion 2026-03-20 (Estimated); Study Completion 2026-03-20 (Estimated)

PRIMARY OUTCOMES:
Ability of PD-L1 to predict response | Up to 3 years
  Based on the results from Part A, the Youden Index methodology will be used to determine the optimal threshold for PD-L1 expression in correlation with tumor response, and if a correlation is identified this threshold will be used for Part B. The overall ability of PD-L1 to predict response will be assessed using the area under the receiver operating characteristic curve (area under the curve). If the area is significantly greater than 0.5, part B will begin using the optimum cutpoint as determined from the Youden index.

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 3 years
  Kaplan-Meier curves will be generated for OS. Median OS will be estimated along with 90% confidence intervals using the method of Brookmeyer and Crowley.
Progression free survival (PFS) | Time from enrollment until disease progression or death from any cause, assessed up to 3 years
  Kaplan-Meier curves will be generated for PFS. Median PFS will be estimated along with 90% confidence intervals using the method of Brookmeyer and Crowley.
Disease control rate (CR + PR + SD) | Up to 3 years
  The disease control rate (CR+PR+SD) and 90% confidence interval will also be determined.

OTHER OUTCOMES:
CD8 TILs will be assessed by percentage of tumor showing infiltration | Baseline
  CD8 levels will be correlated with PD-L1 expression using Pearson or Spearman rank correlation coefficients.
Composite measure of other immune escape mechanisms including MDSCs and other checkpoints | Up to 3 years
  Other immune escape mechanisms including MDSCs and other checkpoints will be assessed by immunohistochemistry (0 - 3+) or flow cytometry counting the number and percentage of positive cells. Levels will be correlated with PD-L1 expression and other biomarkers.
PD-L1 expression by mass spectrometry | Baseline
  PD-L1 expression by mass spectrometry and correlation with PD-L1 expression by IHC as well as tumor response, and the T-cell inflamed phenotype will be performed. Multivariate logistic regression will be performed to determine whether these biomarkers or combinations of biomarkers are predictive of response. Exact logistic regression models will be fit given the small number of responders expected (4 from part A and 7-8 from part B).
Mass spectrometry-based flow cytometric analysis | Up to 3 years
  Mass spectrometry-based flow cytometric analysis (CyTOF) will be descriptive based on number and percentage of certain cell populations.
Analysis of T-cell receptor repertoire from TILs | Up to 3 years
  Analysis of T-cell receptor repertoire from TILs will be descriptive looking for presence or absence of oligoclonal T-cell population.
Duration of response | Up to 3 years
  Will be estimated by Kaplan-Meier.
Incidence of toxicities graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 | Up to 30 days after completion of study treatment
  Toxicities will be summarized in tabular form by type and severity and incidence rates generated.

CONTACTS AND LOCATIONS:
Overall Officials: Hedy Kindler, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States